CLINICAL TRIAL: NCT01323036
Title: Assessment of Bioavailability of Krill Oil Compared to Fish Oil in Healthy Volunteers
Brief Title: Krill Oil Study Compared to Fish Oil
Acronym: Krill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Enzymotec (Industry)
Responsible Party: Principal Investigator, Dr. Peter Jones, Director of RCFFN, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2011:014
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Krill Oil (Experimental)
  Interventions: Dietary Supplement: Krill oil
- Fish Oil (Experimental)
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Krill oil — Krill oil:Total omega-3 fatty acids: 560-660 mg and Astaxanthin: 1800 µg
  Arms: Krill Oil
Dietary Supplement: Fish Oil — Fish oil: Total omega-3 fatty acids: 560-660 mg
  Arms: Fish Oil

SUMMARY:
The main purpose of the study is to evaluate the absorption of omega-3 fatty acids into the blood following consumption of krill oil compared with fish oil and placebo.

DETAILED DESCRIPTION:
The main purpose of the study is to evaluate the absorption of omega-3 fatty acids into the blood following consumption of krill oil compared with fish oil and placebo. An additional purpose is to evaluate the lipid-lowering efficacy and safety of consumption of Krill Oil and Fish Oil to a placebo product. It has been shown that the ingestion of Krill Oil leads to better absorption of omega-3 fatty acids compared to ingestion of Fish Oil. It was also shown that consumption of krill oil and fish oil result in a favorable modification of lipid profiles. Therefore, it is anticipated that consumption of these krill oil and fish oil will improve lipid profile, as well as other health-related markers and will be safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and premenopausal not pregnant or nursing women between 18 and 49 years old.

Exclusion Criteria:

* smokers
* rheumatoid arthritis
* chronic illness
* cardiovascular problems
* dyslipidemia
* liver and kidney disease
* diabetes
* endocrine or metabolic disease
* inflammatory bowel disease
* pancreatitis
* gallbladder or biliary disease
* neurological/psychological disease
* bleeding disorders
* experienced platelet abnormalities
* gastrointestinal disorders that could interfere with fat absorption
* hypertension
* history of cancer
* an intention to lose weight
* use of anticoagulant
* serum triglycerides (TG) >200 mg/dL, and/or total cholesterol (TC) >240 mg/dL, and/or LDL-cholesterol (LDL-C) >160 mg/dL
* hypertension or lipid lowering medications
* consumption of more than one alcoholic drinks/day
* Consumption of more than one fish or seafood serving
* one month prior to the start of the study
* omega-6 fatty acids in the past 6 months
* planned to consume seafood products or fish or to use any omega-3 or omega-6 fatty acids nutritional supplements at anytime in the duration of the study
* planned to to become pregnant during the study period
* BMI>28
* allergies to fish seafood or corn

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Ramprasath VR, Eyal I, Zchut S, Shafat I, Jones PJ. Supplementation of krill oil with high phospholipid content increases sum of EPA and DHA in erythrocytes compared with low phospholipid krill oil. Lipids Health Dis. 2015 Nov 4;14:142. doi: 10.1186/s12944-015-0142-y. PMID 26537218
- [Derived] Ramprasath VR, Eyal I, Zchut S, Jones PJ. Enhanced increase of omega-3 index in healthy individuals with response to 4-week n-3 fatty acid supplementation from krill oil versus fish oil. Lipids Health Dis. 2013 Dec 5;12:178. doi: 10.1186/1476-511X-12-178. PMID 24304605